CLINICAL TRIAL: NCT05920694
Title: Restoring Metabolic and Reproductive Health With Sleep in PCOS Study, CPAP Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-36861
Record Dates: First submitted 2023-06-05; First posted 2023-06-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovary Syndrome; Obstructive Sleep Apnea
MeSH Terms: conditions — Polycystic Ovary Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CPAP Group (Active Comparator): Participants randomized to CPAP will initiate CPAP therapy at the beginning of the study.
  Interventions: Device: Continuous Positive Airway Pressure Device (CPAP)
- Delayed CPAP Group (Placebo Comparator): Participants randomized to delayed CPAP (waitlist control) will initiate CPAP therapy immediately after 12 weeks. The investigators recognize that adherence to CPAP therapy is a common barrier to effective clinical treatment of OSA and to rigorous research on CPAP and has been significantly correlated with improvements in insulin resistance, including in a small of study of women with PCOS. After receiving this device, participants can meet with a study psychiatrist and his team within 3 days of initiating CPAP therapy and as needed for up to a month after initiating therapy. No visits in this time period will be billed to insurance.
  Interventions: Other: Delayed Continuous Positive Airway Pressure Device (CPAP)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure Device (CPAP) — Metabolic studies will be performed before and after initiation of CPAP therapy, which is currently the first-line standard of care for treatment of patients with OSA, both with and without hypoxia.
  Arms: CPAP Group
Other: Delayed Continuous Positive Airway Pressure Device (CPAP) — Metabolic studies will be performed before and after the study period of 12 weeks. After 12 weeks, participants will immediate receive CPAP therapy, which is currently the first-line standard of care for treatment of patients with OSA, both with and without hypoxia.
  Arms: Delayed CPAP Group

SUMMARY:
In this study, the researchers are trying to learn more about the relationship between Polycystic Ovary Syndrome and Obstructive Sleep Apnea (OSA). Obstructive Sleep Apnea is a sleep-related breathing disorder that involves a decrease or complete stop in airflow. The purpose of this study is to find out why some people with obstructive sleep apnea have higher levels of insulin resistance, and the investigators will study the role of hypoxia (low levels of oxygen in the blood at night) in insulin resistance and see if insulin resistance improves during your treatment with CPAP.

DETAILED DESCRIPTION:
Today, approximately 5 million Americans of reproductive age have Polycystic Ovary Syndrome (PCOS). The personal and public health burden of PCOS is high. People with PCOS are at elevated risk of infertility, endometrial cancer, obesity, diabetes, dyslipidemia and nonalcoholic fatty liver disease (NAFLD). Moreover, there is a paucity of treatments that address the metabolic and reproductive concerns of this disorder. Obstructive sleep apnea (OSA) is a recognized co-morbidity of PCOS that may exacerbate both metabolic and reproductive aspects of PCOS. Thus, treating OSA represents a potentially attractive tool to improve outcomes in PCOS. Indeed, continuous positive airway pressure therapy (CPAP) is a relatively inexpensive treatment for OSA that is safe for use in women in the reproductive years, even when pregnant or trying to conceive. However, evidence regarding the impact of CPAP use in PCOS populations is lacking, and, currently, screening and treatment of OSA is only considered standard of care to treat symptoms of excessive sleepiness or hypertension. Because an estimated 15-45% of people with moderate/severe OSA do not have these symptoms, treatment is not considered standard of care for the majority of persons with OSA and PCOS. From another study looking at sleep and PCOS, we will identify 20 subjects with moderate-to-severe OSA without excessive daytime sleepiness who will enroll in a CPAP trial. These subjects will undergo intensive multi-tissue insulin resistance testing and will be assigned treatment with CPAP or delayed treatment after 12 weeks after which all measures will be re-assessed. Accordingly, this proposal will address an unanswered question: Does CPAP provide metabolic or reproductive benefits in PCOS? The results will also better define potential mechanistic pathways linking OSA to insulin resistance and will determine whether CPAP improves key outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects found to have moderate to severe OSA (AHI >15)
* PCOS diagnosis satisfies both the hyperandrogenic and oligo-ovulatory requirements of Rotterdam criteria
* Ages 18-40
* BMI 25-45 kg/m2
* Fasting insulin >16
* At-risk score on Berlin Questionnaire

Exclusion Criteria:

* Current use of oral contraceptives
* Diabetes mellitus (fasting glucose ≥126 mg/dL or 2-h glucose ≥200 mg/dL or HGB A1c ≥6.5%)
* Treatment for asthma
* Regular tobacco use or alcohol consumption exceeding 1 drink/day
* HIV infection or infectious hepatitis
* Pregnancy or lactation within the past six months
* Prior OSA treatment
* Excessive daytime sleepiness as defined as >16 on the Eppworth Sleepiness Scale or untreated or inadequately treated hypertension (>150/90)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants showing a change in fractional de novo lipogenesis (DNL, %) | Baseline and 12 weeks
  The percent of newly synthesized fatty acids (DNL, %) will be measured using a stable isotope (deuterated water) and mass spectrometry.
Number of participants showing a change in free testosterone (pg/mL) | Baseline and 12 weeks
  The aim is evaluate the effect of treating OSA with CPAP on biochemical hyperandrogenism in individuals with PCOS.
Number of participants showing a change in insulin secretion rate (picomol/min) | Baseline and 12 weeks
  Glucose Tolerance Test is used to measure of insulin secretion rate.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No